CLINICAL TRIAL: NCT06425172
Title: A Monitoring System for Cranial Remolding Orthoses
Brief Title: Monitoring System for Cranial Orthoses
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tiffany Graham, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2022-0556
Record Dates: First submitted 2024-04-30; First posted 2024-05-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Plagiocephaly; Brachycephaly; Deformational Plagiocephaly; Deformational Posterior Plagiocephaly
MeSH Terms: conditions — Plagiocephaly; Craniosynostoses; Plagiocephaly, Nonsynostotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Infants with with deformational head shapes: Infants who have been referred for custom orthotic treatment for a deformational head shape such as deformational plagiocephaly or deformational brachycephaly.
  Interventions: Device: Cranial Remolding Orthosis

INTERVENTIONS:
Device: Cranial Remolding Orthosis — A custom made FDA-approved cranial remolding orthosis will be retrofit with sensors used in the research.
  Other Names: Custom Helmet

SUMMARY:
This is a study which investigates the wear time and fit of a cranial remolding orthosis (a standard-of-care treatment where an infant wears a custom helmet to help reshape their head as they grow).

DETAILED DESCRIPTION:
This is a study which investigates the wear time and fit of a cranial remolding orthosis (a standard-of-care treatment where an infant wears a custom helmet to help reshape their head as they grow). Although cranial remolding treatment has been used successfully for over 20 years, there is no clinical standard for objective monitoring of the fit and wear time.

In total, participation will consist of 7 visits over 11 weeks: (1) measurements and clinical evaluation [approximately 60 minutes], (2) fitting of standard helmet and pre-fitting and/or fitting of the research helmet [approximately 60 minutes], (3) fitting of research helmet (if not done at Visit #2) and in-office testing [approximately 2 hours], (4)/(5)/(6) follow up visits for research helmet [approximately 30-60 minutes each], and (7) final follow up visit and in-office testing for the research helmet [approximately 2 hours].

During the 8-9 weeks of wearing the research helmet, the child is expected to wear the it 23 hours per day (after a break-in schedule), and caregivers will keep a log of helmet wear time and any side effects (such as skin irritations), if they occur. The child will be seen clinically every 2 weeks (or more often, if caregivers request additional checkups).

At the end of the trial, participants will return all research-related materials and the treating clinician will return the child to wearing the standard helmet.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are clinically indicated for cranial remolding orthoses for treatment of a deformational head shape (i.e. plagiocephaly / brachycephaly)

Exclusion Criteria:

* non-English speaking caregivers
* infants with craniosynostosis or those not indicated for cranial remolding
* infants with developmental comorbidities which affect cranial growth

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants who are clinically indicated for cranial remolding orthoses.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Wear time monitoring and validation | Data will be recorded for 8-9 weeks per subject, and analyzed throughout the study. Anticipated to be complete on all subjects within 1 year.
  The temperature readings from the custom temperature sensor within the research helmet will be compared to the collected temperature readings from the iButtons. Using established software compatible with the iButton, wear time will be calculated based on previously reported temperature thresholds which indicate the helmet is being worn. Using similar temperature thresholds, wear time data from the custom sensors will be compared to the wear time reported by the iButton software.
Fit monitoring | Data will be recorded for 8-9 weeks per subject, and analyzed throughout the study. Anticipated to be complete on all subjects within 1 year.
  The investigators will examine pressure in the void space of the helmet throughout the 8-9 weeks of wear time. In theory, the pressure in this area should never increase as the cranium should not come in contact with this sensor no matter what position the infant is in (i.e. laying down, sitting, etc).

SECONDARY OUTCOMES:
Survey Participation | Survey to be taken at completion of the study, anticipated to be complete on all subjects within 1 year.
  Parents will take a survey regarding their experience with the research helmet
Wear time comparison between objective and subjective reporting | Data will be recorded for 8-9 weeks per subject, and analyzed throughout the study. Anticipated to be complete on all subjects within 1 year.
  The wear time based on iButton and custom temperature readings will be compared to the caregiver-reported wear time log and any differences in log times reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Graham, MS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be protected and only shared within the research team and treating practitioners.